CLINICAL TRIAL: NCT03233646
Title: Evaluating the Retinal and Choroidal Microvasculature and Structure Using Multimodal Retinal and Choroidal Imaging in Neurodegenerative Disease: iMIND Research Study
Brief Title: Retinal Imaging in Neurodegenerative Disease
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of Edinburgh in Scotland (Unknown); Tan Tock Seng Hospital in Singapore (Unknown); Queens University of Belfast United Kingdom (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00111831
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment; Parkinson's Disease; Multiple Sclerosis; Huntington Disease; Lewy Body Dementia; Frontotemporal Dementia; Amyotrophic Lateral Sclerosis (ALS); APOE-4 Positive; Traumatic Brain Injury; Concussion; Post-Traumatic Stress Disorder; Down Syndrome; Neuro-Degenerative Disease; Normal Cognition
Keywords: OCT angiography (OCTA); Optical Coherence Tomography (OCT); Vessel Density; Superficial Capillary Plexus; Retinal microvasculature; Scanning Laser Ophthalmoscopy; Ultra-widefield (UWF) Imaging; Perfusion Density; Retinal Nerve Fiber Layer; Ganglion Cell Inner Plexiform Layer; Choroidal Vascularity Index
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Parkinson Disease; Multiple Sclerosis; Huntington Disease; Lewy Body Disease; Frontotemporal Dementia; Amyotrophic Lateral Sclerosis; Brain Injuries, Traumatic; Brain Concussion; Stress Disorders, Post-Traumatic; Down Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Case: Patients with (MCI, PD, AD, FTD, DLB, ALS, MS, HD, TBI, concussion, PTSD and other neurodegenerations as well as Down Syndrome)
  Interventions: Device: Retinal and Choroidal Imaging
- Controls: Controls will be recruited from the relatives/attendants of study participants or will be patients themselves and will not have a neurodegenerative disease diagnosis.
  Interventions: Device: Retinal and Choroidal Imaging

INTERVENTIONS:
Device: Retinal and Choroidal Imaging — Non-invasive OCT, OCTA, and UWF fundus photography of retina

SUMMARY:
This study aims to develop and evaluate biomarkers using non-invasive optical coherence tomography (OCT) and OCT angiography (OCTA) as well as ultra-widefield (UWF) fundus photography to assess the structure and function of the retinal and choroidal microvasculature and structure in persons with mild cognitive impairment (MCI) and Alzheimer's Disease (AD), Parkinson's Disease (PD), or other neurodegenerative disease, diseases as outlined.

DETAILED DESCRIPTION:
Using a multidisciplinary approach, this study aims to yield new insight into the vascular and structural pathophysiology of neurodegenerative disease. The investigators propose to develop and evaluate imaging biomarkers from OCT, OCTA, and UWF fundus photos to assess the structure and function of the retinal and choroidal microvasculature and structure in these individuals.

The investigators hypothesize that microvascular and structural network alterations in the retina and choroid may mirror and possibly precede changes in the cerebral microcirculation seen in these neurodegenerative diseases. Using advanced image analysis and machine learning techniques, the investigators aim to evaluate markers of reduced capillary blood flow and non-perfusion in the superficial retinal vascular plexus and choriocapillaris imaged using OCT and OCTA, in a resolution not previously possible, that would complement already established retinal structural markers and increase their sensitivity and specificity in the earlier detection of these neurodegenerative diseases.

This study looks to provide a proof of concept for retinal and choroidal imaging-based microvascular and structural biomarkers as an effective screening tool for neurodegenerative disease, particularly during in cognitive aging.

The protocol for this study was amended and the record was updated accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Adults with neurodegenerative disease ((MCI, PD, AD, FTD, DLB, ALS, MS, HD, TBI, concussion, PTSD and other neurodegenerations as well as Down Syndrome)
* Adults without neurodegenerative disease

Exclusion Criteria:

* Inability to cooperate with or complete testing or other neurologic or age- related ocular conditions that would impact image acquisition.
* Eyes that have had intraocular surgery, other than cataract surgery.

If two eyes satisfy the inclusion criteria, both eyes will be included in the study. If one eye satisfies the inclusion criteria, the eye that qualifies will be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurology Clinics and the community.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in ganglion cell-inner plexiform layer (GCIPL) thickness | Baseline, 1 year
  Ganglion cell inner plexiform layer thickness as measured on optical coherence tomography scan of macula
Change in retinal nerve fiber layer (RNFL) thickness | Baseline, 1 year
  Retinal nerve fiber layer thickness as measured on optical coherence tomography scan of macula
Change in central subfield thickness (CST) | Baseline, 1 year
  Central subfield thickness as measured on optical coherence tomography scan of macula
Change in choroidal vascularity index (CVI) | Baseline, 1 year
  Choroidal vascularity index as measured using the COIN software in 1500 um area centered on the fovea
Change in foveal avascular zone (FAZ) area | Baseline, 1 year
  Foveal avascular zone area as measured in the superficial capillary plexus on 3mm optical coherence tomography angiography scan of the macula
Change in average perfusion density (PD) | Baseline, 1 year
  Average perfusion density as measured in the ETDRS 3mm and 6mm circle and rings on optical coherence tomography angiography scan of the macula
Change in average vessel density (VD) | Baseline, 1 year
  Average vessel density as measured in the ETDRS 3mm and 6mm circle and rings on optical coherence tomography angiography scan of the macula
Change in average capillary perfusion density (CPD) | Baseline, 1 year
  Capillary perfusion density as measured on peripapillary 4.5mm optical coherence tomography angiography scan
Change in average capillary flux index (CFI) | Baseline, 1 year
  Capillary flux index as measured on peripapillary 4.5mm optical coherence tomography angiography scan

SECONDARY OUTCOMES:
Change in retinal vessel tortuosity | Baseline, 1 year
  Retinal vessel tortuosity measured on ultra-widefield scanning laser ophthalmoscopy image using VAMPIRE software
Change in retinal vessel width gradient | Baseline, 1 year
  Retinal vessel width gradient measured on ultra-widefield scanning laser ophthalmoscopy image using VAMPIRE software
Change in retinal vessel fractal dimension | Baseline, 1 year
  Retinal vessel fractal dimension measured on ultra-widefield scanning laser ophthalmoscopy image using VAMPIRE software

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Fekrat, MD FACS FASRS, Principal Investigator — Duke University; Dilraj Grewal, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao W, Robbins CB, Grewal DS, Patel H, Soundararajan S, Liu AJ, Johnson KG, Agrawal R, Petrella JR, Stinnett SS, Parker D, Fekrat S. Correlating retinal and choroidal vascular parameters with volumetric MRI in Alzheimer's disease and amnestic mild cognitive impairment. BMC Ophthalmol. 2025 Jul 1;25(1):365. doi: 10.1186/s12886-025-04157-x. PMID 40598011
- [Derived] Robbins CB, Akrobetu D, Ma JP, Stinnett SS, Soundararajan S, Liu AJ, Johnson KG, Grewal DS, Fekrat S. ASSESSMENT OF RETINAL MICROVASCULAR ALTERATIONS IN INDIVIDUALS WITH AMNESTIC AND NONAMNESTIC MILD COGNITIVE IMPAIRMENT USING OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY. Retina. 2022 Jul 1;42(7):1338-1346. doi: 10.1097/IAE.0000000000003458. PMID 35723922